CLINICAL TRIAL: NCT04237675
Title: Assessment of Risk of Postoperative Relapses in Patients With Multiple Sclerosis; an Observational Study
Brief Title: Postoperative Relapses in MS Patients
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Staikou Chryssoula, Associate Professor, University of Athens
Other Study IDs: 157/19-12-19
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis Relapse; Surgery; Anesthesia
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- regional anesthesia
  Interventions: Procedure: surgery and anesthesia
- general anesthesia
  Interventions: Procedure: surgery and anesthesia

INTERVENTIONS:
Procedure: surgery and anesthesia — patients with MS who received general or regional anesthesia for a surgery or labor

SUMMARY:
The aim of the study is to record any relapses during one year postoperatively in patients and parturients diagnosed with MS who received general or regional anesthesia

ELIGIBILITY:
Inclusion Criteria: diagnosed MS -

Exclusion Criteria: refuse to participate

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients or parturients with MS who received general or regional anesthesia for surgery or labor analgesia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MS relapses | one year postoperatively
  number of relapses

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Aretaieio Hospital, University of Athens, Athens, Attica
  - Aretaieio Hospital, Athens

IPD SHARING:
Plan to Share IPD: Undecided